CLINICAL TRIAL: NCT02761824
Title: Implementation and Evaluation of an Activity Based Program to Improve Quality of Life Outcomes in Women Diagnosed With Cancer
Brief Title: Activity Based Program to Improve Quality of Life Outcomes in Women Diagnosed With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Sciences in Philadelphia (Other)
Collaborators: Temple University (Other); M.D. Anderson Cancer Center (Other); Dolfinger-McMahon Foundation (Unknown); Genesis Health System (Other)
Responsible Party: Principal Investigator, Colleen Maher, Primary Investigator, University of the Sciences in Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 342186-7
Record Dates: First submitted 2016-04-29; First posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Cancer
Keywords: Quality of Life; Occupation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Camp Discovery (Experimental): One week activity based camp.
  Interventions: Other: Camp Discovery

INTERVENTIONS:
Other: Camp Discovery — Activities included physical, social, emotional, sensory and spiritual activities.

SUMMARY:
Implementation and Evaluation of an Activity Based Program to Improve Quality of Life Outcomes in Women Diagnosed With Cancer. Demonstrate improved life satisfaction (with evidenced gathered at three consecutive periods and geographical locations through Quality of Life surveys).

DETAILED DESCRIPTION:
This research study focused on developing and implementing eight one-week activity camps in the summer of 2012, 2013, and 2014 for women diagnosed with cancer. Each camp was held in a different geographical location: rural (Renovo, PA), suburban (Gilda's Club in Warminster, PA), MD Anderson of Camden, and urban (University of the Sciences with the Cancer Support Community of Philadelphia). The focus of this programming was to allow women to engage in activities they may not be engaged in since the diagnosis of cancer and to provide them with opportunities to socially interact and communicate with individuals who may have encountered the same difficulties as them. Quality of life information was collected before, during and after implementation of the activity program. The main objective was to demonstrate improved life satisfaction (with evidenced gathered at three consecutive periods and geographical locations through Quality of Life surveys). 77 women were recruited over a three year period. 6 dropped out and 71 completed the entire study.

ELIGIBILITY:
Inclusion Criteria:

* women diagnosed with cancer
* age of 21 or older
* a clearance from their MD to participate in the activity program.

Exclusion Criteria: Not Applicable (NA)

* none

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in Canadian Occupational Performance Measure Scores at Day 5 and Week 6 | Day 1, Day 5 and week 6
  Individualized, client-centered measure designed for use by occupational therapists to detect change in a client's self-perception of occupational performance and satisfaction over time
Change in World Health Organization-Quality of Life Brief (WHO-QoL BREF )scores at Week 6 | Day 1 and week 6
  Quality of Life Measure: Assesses the individual's perceptions in the context of their culture and value systems, and their personal goals, standards and concerns.
Change in Short Form 36 (SF 36) at Week 6 | Day 1 and week 6
  Multi-purpose, short-form health survey with 36 questions. Yields a profile of functional health and well-being scores. Provides psychometrically based physical and mental health summary measures.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen M Maher, OTD, Principal Investigator — University of Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maher C, Mendonca RJ. Impact of an Activity-Based Program on Health, Quality of Life, and Occupational Performance of Women Diagnosed With Cancer. Am J Occup Ther. 2018 Mar/Apr;72(2):7202205040p1-7202205040p8. doi: 10.5014/ajot.2018.023663. PMID 29426382